CLINICAL TRIAL: NCT05424757
Title: Quantitative Analysis of Selected PEG 3350 Components and Metabolites in Children's Plasma and Urine
Brief Title: Polyethylene Glycol Safety in Children
Status: Completed | Type: Observational
Sponsor: Children's Hospital of Philadelphia (Other)
Collaborators: Food and Drug Administration (FDA) (U.S. Federal Agency)
Responsible Party: Sponsor
Other Study IDs: 14-011454; 1R01FD005312-01 (FDA)
Record Dates: First submitted 2022-06-15; First posted 2022-06-21 (Actual); Last update posted 2025-11-04 (Actual); Status verified 2025-11

CONDITIONS: Polyethylene Glycols; Children, Only
MeSH Terms: interventions — polyethylene glycol 3350

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Cross-Sectional
Patient Registry: Yes
Target Follow-Up Duration: 1 Day
Biospecimen Retention: Samples Without DNA — * Blood: 1.5 mL (up to 6 months of age), 2.5 mL (6 to 24 months old), 5 mL (older than 24 months). No more than 3 mL/kg will be collected from any child.
  * Urine (10 mL)
  * Stool (10-20 grams for possible future analyses)
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

GROUPS / COHORTS (2):
- Children who are taking PEG 3350: * Children less than 17 years old who have taken PEG 3350 daily for at least 30 days.
  * Dose of PEG 3350 greater than or equal to 0.4 grams/kg/day.
  * Preference will be given to children taking at least 17 grams/day.
  Notes:
  Only children who are already taking PEG 3350 as part of their current medical regimen will be included. Changes to medical therapy are not recommended as part of this study.
  Children in three subgroups will be enrolled:
  1. Children with no known bowel or nervous system disease or neuropsychiatric symptoms.
  2. Children with bowel problems that might increase intestinal permeability.
  3. Children with neurologic disease or with neuropsychiatric disorders or symptoms.
  Interventions: Drug: PEG 3350
- Children who are not taking PEG 3350: * Children less than 17 years old who have NOT taken PEG 3350 for at least 30 days.
  Children in three subgroups will be included:
  1. Children with no known bowel or nervous system disease or neuropsychiatric symptoms.
  2. Children with bowel problems that might increase intestinal permeability.
  3. Children with neurologic disease or with neuropsychiatric disorders or symptoms.

INTERVENTIONS:
Drug: PEG 3350 — Data and biospecimens will be collected from two groups of children:
  * Children who have taken PEG 3350 daily for at least 30 days.
  * Children who have NOT taken PEG 3350 for at least 30 days.
  No changes to medicines are recommended as part of this study.
  Groups: Children who are taking PEG 3350

SUMMARY:
The primary objective is to measure levels of selected PEG 3350 components and metabolites in the blood and urine of children who are already taking PEG 3350 compared to children who are not taking PEG 3350.

Changes to medical therapy are not recommended as part of this study.

DETAILED DESCRIPTION:
For subjects taking PEG 3350, blood and urine will be collected 1.5 to 4 hours after subjects take PEG 3350.

For subjects who are not taking PEG 3350, the same PEG 3350 components and metabolites will be measured in blood and urine.

PEG 3350 containing medicines from study subjects will be analyzed for the same PEG 3350 components and metabolites.

A stool specimen will be collected for future studies.

Additional data will be obtained from:

* Review of medical records.
* A brief questionnaire.
* Child Behavior Checklist (CBCL) from the Achenbach System of Empirically Based Assessment (for children more than 1.5 years old)
* Bayley-IV Social-Emotional Scale assessment (for children less than 1.5 years old)

ELIGIBILITY:
Group 1: Children who do not have bowel or nervous system disease, or neuropsychiatric symptoms.

Inclusion criteria:

Children less than 17 years old who have been taking PEG 3350 for at least one month.

Dose of PEG 3350 greater than or equal to 0.4 grams/kg/day currently recommended by the North American Society for Pediatric Gastroenterology, Hepatology and Nutrition (NASPGHAN) and European Society for Pediatric Gastroenterology, Hepatology and Nutrition (ESPGHAN) guidelines (2). Preferences will be given to children taking at least 17 grams/day.

Normal Physical and neurological development for age. Weight and height percentiles ≥ 5% and ≤ 95% for age.

Exclusion criteria:

Children with underlying bowel problems that might be expected to increase bowel permeability (are included in group 2). In this group we will specifically exclude children with:

Diarrhea within the past month. Note that PEG 3350 may cause loose stool and this is often the intended therapeutic effect. Therefore, we will exclude children with presumed infectious diarrhea since this may alter gut permeability but will include children whose loose stool is attributed to PEG 3350. If loose or watery stool began after initiation of PEG 3350 or after an increase in PEG 3350 dose within prior 3 days, children may be enrolled for GROUP 1.

Children whose stool had a recognized diarrhea causing pathogen within the past 4 months will be excluded since the time required to repair epithelial lining is not clear. Enteric pathogens that would prevent enrollment include Salmonella, Shigella, Campylobacter, Yersinia, E. Coli (enterotoxigenic, enteropathogenic, enteraggregative, enterohemorrhagic), Clostridum difficile, Rotavirus, Norovirus, Astrovirus, and other known or suspected diarrhea causing organisms.

H. pylori infection since this causes a stomach inflammation. HIV infection since this may alter bowel permeability (17) and predispose to other types of infection Symptoms neurologic disease or dysfunction (since they will be enrolled in Group 3).

Group 2: Children with problems that might increase intestinal epithelial permeability.

Inclusion criteria:

Children less than 17 years old who have been taking PEG 3350 for at least one month.

Dose of PEG 3350 greater than or equal to 0.4 grams/kg/day currently recommended by the NASPGHAN and ESPGHAN guidelines (2). Preferences will be given to children taking at 17 grams/day.

c. Any of the following problems associated with increased bowel permeability:

* Weight ≤ 5% for age. Malnutrition is associated with increased intestinal permeability.
* Children who had a pathogen (see Group 1 Exclusion Criteria "A. b." for list of pathogens) isolated from their stool within the past month.
* Children with celiac disease who are untreated or began treatment within the past 3 months.
* Children with inflammatory bowel disease
* Children with Hirschsprung disease. This intestinal motility disorder predisposes to bowel injury called enterocolitis (18-20).
* Children with intestinal motility disorders other than Hirschsprung disease.

Exclusion criteria:

a. Children with neurologic or neuropsychiatric symptoms. These children will be enrolled in Group 3.

Group 3: Children with underlying neurologic disease or with neuropsychiatric disorders or symptoms.

Inclusion criteria:

Children less than 17 years old who have been taking PEG 3350 for at least one month.

Dose of PEG 3350 greater than or equal to 0.4 grams/kg/day currently recommended by the NASPGHAN and ESPGHAN guidelines (2). Preference will be given to children taking at least 17 grams/day.

Any of the following problems with the nervous system:

* Diagnosed with a disease that affects nervous system function before starting PEG 3350.
* Diagnosed with a disease that affects nervous system function after starting PEG 3350.
* Abnormal nervous system function without a specific diagnosis.
* Episodic nervous system dysfunction. This might include seizure disorder, metabolic disease, or mitochondrial disease.

Note: Included in Group 3 are children with cerebral palsy, neuronal migration defects, traumatic brain injury, hypoxic ischemic encephalopathy, seizure disorder, tics, migraine, clinical depression, anxiety disorder, obsessive-compulsive disorder, post-surgical brain injury, autism spectrum disorder as well as genetic defects that affect the nervous system (Cornelia de Lange, Rett Syndrome, Pelizaeus-Merzbacher disease, etc.).

Any weight and height (i.e., no exclusions based on growth percentiles). Abnormalities in any organ including the bowel are acceptable.

Exclusion criteria:

a. There are no specific exclusion criteria. This is important since this group may be at the highest risk for PEG 3350 side effects.

Group 4: Children who are not taking PEG 3350. We will enroll 75 children who are not taking PEG 3350. Inclusion and exclusion criteria for these children will be the same as those detailed above for children who are taking PEG 3350 except that they may not have taken PEG 3350 within the last month.

Enrollment targets for Groups 1, 2 and 3:

1. 15 children taking PEG 3350, age 0-6 years old (for each Group).
2. 6 children taking PEG 3350, age 7-12 years old (for each Group).
3. 4 children taking PEG 3350, age 13-17 years old (for each Group).
4. An equal number of children in each age group who are not taking PEG 3350.

Ages: 0 Years to 16 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Study Population: Study population will be selected from children cared for at The Children's Hospital of Philadelphia.
Sampling Method: Non-Probability Sample
Enrollment: 158 (Actual)
Dates: Start 2022-09-30 (Actual); Primary Completion 2025-08-09 (Actual); Study Completion 2025-08-09 (Actual)

PRIMARY OUTCOMES:
PEG 3350 related molecules in plasma | 15 minutes
  Plasma levels of selected PEG 3350 related molecules will be measured by mass spectrometry using validated assays.
PEG 3350 related molecules in urine | 10 minutes
  Urine levels of selected PEG 3350 related molecules will be measured by mass spectrometry using validated assays.
PEG 3350 related molecules in medicine samples | 5 minutes
  Medicine sample levels of selected PEG 3350 related molecules will be measured by mass spectrometry using validated assays.
Neurobehavioral symptoms in children who are taking PEG 3350 | 5 minutes
  Participants will complete a short symptom questionnaire specific to this study. The questionnaire asks if specific symptoms are present and if they changed after the child started PEG 3350 containing medicine.
Baseline neurobehavioral symptoms in children who are not taking PEG 3350 | 5 minutes
  Participants will complete a short symptom questionnaire specific to this study.
Assessment of current Child behavior (1.5 years to 18 years old) | 30 minutes
  Families with children >1.5 years to 18 years old will complete an age-appropriate Child Behavior Checklist (CBCL) from the Achenbach System of Empirically Based Assessment. Specific CBCL forms are available for ages 1.5 to 5 years and for 6 to 18 years.
  Standard scores are scaled. 50 is average for age and gender. Standard deviation is 10 points. Higher scores indicate greater problems. Normal = below 93%. Borderline = 93-97%. Clinical range = above 97%.
Assessment of current Child behavior (< 1.5 years old) | 90 minutes
  Caregivers with children < 1.5 years old will complete a Bayley-4 Social-Emotional Scale (BSID-IV) assessment. The BSID-IV Social-Emotional Scale is an adaptation of the Greenspan Social-Emotional Growth Chart: A Screening Questionnaire for Infants and Young Children. The Social-Emotional Scale assesses acquisition of social and emotional milestones.
  Items assess mastery of functional emotional skills, such as self-regulation and interest in the world; communicating needs; engaging others and establishing relationships; using emotions in a purposeful manner; and using emotional signals to solve problems.
  The standardized mean motor score is 100 (SD 15), with scores lower than 85 indicating mild impairment, and lower than 70 indicating moderate or severe impairment.

CONTACTS AND LOCATIONS:
Overall Officials: Robert O Heuckeroth, MD, PhD, Principal Investigator — Children's Hospital of Philadelphia
Locations (1):
- Children's Hospital of Philadelphia, Philadelphia, Pennsylvania, United States

IPD SHARING:
Plan to Share IPD: No
There is no plan to make individual participant data available to other researchers.